CLINICAL TRIAL: NCT04677816
Title: Impact of Vitamin D Supplementation on the Rate of Pathologic Complete Response in Vitamin D Deficient Patients Receiving Neoadjuvant Chemotherapy for Operable Triple Negative Breast Cancer
Brief Title: Impact of Vitamin D Supplementation on the Rate of Pathologic Complete Response in Vitamin D Deficient Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00074154; WFBCCC 98121 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Triple Negative Breast Cancer; Vitamin D Deficiency; Invasive Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D Supplementation Group - Deficient Levels (Experimental): Along with standard of care neoadjuvant chemotherapy treatments and procedures, participants will receive oral 50,000 international units of Vitamin D3 supplementation at the initiation of chemotherapy once a week.
  Interventions: Drug: Standard of Care Neoadjuvant Chemotherapy (NAC); Dietary Supplement: Vitamin D3; Other: Drug Diary
- Observational Arm - Vitamin D at Normal Levels (Active Comparator): Standard of care neoadjuvant chemotherapy
  Interventions: Drug: Standard of Care Neoadjuvant Chemotherapy (NAC)

INTERVENTIONS:
Drug: Standard of Care Neoadjuvant Chemotherapy (NAC) — Participants will receive standard of care neoadjuvant chemotherapy with doxorubicin (60 mg/m2) and cyclophosphamide (600 mg/m2) for 4 cycles and paclitaxel (80 mg/m2) weekly for 12 cycles. Doxorubicin and cyclophosphamide (AC) may be administered on a classical every 3 week or dose dense every 2-week (with growth factor support) schedule at the treating physician's discretion. Routine incorporation of carboplatin is not required, however use of carboplatin (AUC 1.5 to 2 weekly or AUC 6 on week 1, 4, 7, and 10) with paclitaxel is allowed at the treating investigator's discretion.
  Upon completion of neoadjuvant chemotherapy, all patients will undergo definitive surgery with either breast conservation or mastectomy with axillary lymph node staging. Type of surgery will be determined by the treating physician.
Dietary Supplement: Vitamin D3 — Participants with deficient levels of vitamin D will receive vitamin D supplementation at the initiation of chemotherapy with 50,000 IU of oral vitamin D3 (cholecalciferol) once a week to be continued for 20 weeks during neoadjuvant chemotherapy.
  Arms: Vitamin D Supplementation Group - Deficient Levels
Other: Drug Diary — Participants that will receive Vitamin D will be asked to fill out a drug diary on a daily basis. Compliance and feasibility will be assessed through a drug diary and pill counts at set time points.
  Arms: Vitamin D Supplementation Group - Deficient Levels

SUMMARY:
A two arm pilot study investigating the rate of pathologic complete response in patients with vitamin D deficiency and triple negative breast cancer undergoing standard neoadjuvant chemotherapy + vitamin D supplementation, including an observational arm to describe response in patients who are not deficient. Investigators hypothesize that vitamin D supplementation during neoadjuvant chemotherapy in operable triple negative breast cancer patients with vitamin D deficiency, will increase the rate of pathologic complete response chain reaction to that of vitamin D sufficient patients based on historical controls.

DETAILED DESCRIPTION:
Primary Objective: To determine if pathologic complete response in vitamin D deficient patients receiving vitamin D supplementation during neoadjuvant chemotherapy for operable triple negative breast cancer is greater than or equal to 60% or less than or equal to pathologic complete response in historical controls (30%) using a one-stage phase II design.

Secondary Objective(s):

* To estimate the proportion of patients with residual cancer burden (RCB) classes I, II, and III in vitamin D deficient patients receiving vitamin D supplementation during neoadjuvant chemotherapy for operable triple negative breast cancer.
* To estimate pathologic complete response reaction in the observational arm of vitamin D sufficient patients receiving neoadjuvant chemotherapy for operable triple negative breast cancer.
* To determine the feasibility of delivery of vitamin D supplementation with standard of care chemotherapy.
* To determine the safety and tolerability of the combination of vitamin D supplementation with standard of care chemotherapy.
* To estimate the change in vitamin D receptor (VDR) expression from pre- and post-neoadjuvant treatment breast tumor tissue samples of vitamin D deficient patients.
* To estimate the change in VDR expression from pre- to post-neoadjuvant treatment breast tumor tissue samples in a sample of 5 vitamin D sufficient patients.
* To estimate the changes in the fecal microbiome and mammary gland microbiome of vitamin D deficient patients from pre- to post-neoadjuvant treatment, and to explore the concordance in the changes between the mammary and fecal microbiome.
* To estimate the changes in the fecal microbiome and mammary gland microbiome in a sample of 5 vitamin D sufficient patients from pre- to post-neoadjuvant treatment.

Patients will be followed for a minimum of 30 days after the last study intervention is administered for adverse events monitoring.

Patients will be followed for 30 days after removal from study or until death, whichever occurs first. Patients removed from study for unacceptable adverse events will be followed until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Women or men with histologically confirmed invasive mammary carcinoma.
* Known triple negative ER/PR/HER2 receptor status as defined by:

  * ER and PR less than or equal to 10% and
  * HER2 negative based on one of the following:
  * IHC 0 or 1+
  * IHC 2+ and FISH negative
  * IHC 2+ and FISH equivocal and no indication for HER2 targeted therapy based on the treating investigators discretion (i.e., HER2: CEP17 ratio < 2.0 or HER2 total copy number <6)
* Patients who plan to undergo neoadjuvant chemotherapy prior to definitive surgical management. Participants are eligible up to 2 weeks after initiating neoadjuvant chemotherapy.
* ECOG performance status of 0, 1 or 2.
* Age ≥ 18.
* The effects of high dose vitamin D on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).

Exclusion Criteria:

* Patients with nephrolithiasis within the past year.
* Patients with known sarcoidosis.
* Patients with corrected calcium >10.5 mg/dL within 30 days prior to initiation of chemotherapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vitamin D.
* Pregnant women are excluded from this study because vitamin D supplementation greater than the recommended daily allowance (RDA) is a pregnancy class C agent with no adequate or well controlled studies in humans.
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with high dose vitamin D (greater than RDA), women who are breastfeeding are excluded from this study.
* Prior treatment for this malignancy including surgery, radiation therapy, chemotherapy, hormonal therapy or investigational agent prior to study entry.
* Patients currently taking Vitamin D at a dose of 50,000 International Units (IU) once weekly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Pathologic Complete Response (pCR) in Vitamin D Supplementation Group | Up to 26 months
  Investigators will determine whether the proportion responding (pCR) is less than or equal to 30% or greater than or equal to 60% using a one-stage phase II design. All participants in the intervention group who are evaluable will be included in the analysis. Pathologic complete response, which is also characterized as residual cancer burden 0, is defined as a final surgical pathologic diagnosis of ypT0 ypN0 or ypTis ypN0.

SECONDARY OUTCOMES:
Number of Participants with Residual Cancer Burden (RCB) Index - Vitamin D Supplementation Group | Up to 26 months
  Five variables are included in the calculation formula. These include: 1) Primary tumor bed area, defined as the largest two dimensions (mms) of the residual tumor bed in the breast (largest tumor bed if multicentric disease), 2) Overall cancer cellularity (as percentage of area), 3) Percentage of cancer that is in situ disease, 4) Number of positive lymph nodes and 5) Diameter of largest metastasis. The calculated residual cancer burden index will be categorized as one of four residual cancer burden classes RCB-0 (pathologic complete response), minimal residual disease (RCB-I), moderate residual disease (RCB-II), or extensive residual disease (RCB-III).
Number of Participants with Residual Cancer Burden (RCB) Index - Observational Arm | Up to 26 months
  Five variables are included in the calculation formula. These include: 1) Primary tumor bed area, defined as the largest two dimensions (mms) of the residual tumor bed in the breast (largest tumor bed if multicentric disease), 2) Overall cancer cellularity (as percentage of area), 3) Percentage of cancer that is in situ disease, 4) Number of positive lymph nodes and 5) Diameter of largest metastasis. The calculated residual cancer burden index will be categorized as one of four residual cancer burden classes RCB-0 (pathologic complete response), minimal residual disease (RCB-I), moderate residual disease (RCB-II), or extensive residual disease (RCB-III).
Feasibility of Delivery of Standard NAC and Vitamin D Supplementation - Accrual Rate | Up to 26 months
  Will be calculated as the number of women who agreed to participate divided by the number of months of recruitment. Estimates and 95% confidence intervals will be calculated for all study participants and for the subset of evaluable participants.
Feasibility of Delivery of Standard NAC and Vitamin D Supplementation - Participation Rate | Up to 26 months
  Will be calculated as the percent of eligible participants who agreed to participate. Estimates and 95% confidence intervals will be calculated for all study participants and for the subset of evaluable participants.
Feasibility of Delivery of Standard NAC and Vitamin D Supplementation - Retention Rate | Up to 26 months
  Will be calculated as the number of participants on whom investigators can obtain the final surgery pathology report by the number who consented to participate. Estimates and 95% confidence intervals will be calculated for all study participants and for the subset of evaluable participants.
Feasibility of Delivery of Standard NAC and Vitamin D Supplementation - Adherence Rate | Up to 26 months
  Will be defined by the proportion of Vitamin D supplements consumed and the proportion of women who took at least 80% of pills. Estimates and 95% confidence intervals will be calculated for all study participants and for the subset of evaluable participants.
Number of Adverse Events | Up to 26 months
  To determine safety of intervention all adverse events will be documented and analyzed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 for adverse event reporting using frequencies of events, grade and attribution.
Change in Vitamin D Receptor (VDR) Expression | Up to 26 months
  Investigators will use a paired t-test to examine the change in Vitamin D receptor expression from pre-post neoadjuvant treatment.
Change in Fecal Microbiomes | Up to 26 months
  Investigators will examine the proportion of different bacteria taxa at each time point, and will use a marginalized two-part beta regression model to account for the compositional nature of the data. A list of all the microbiologic species will be recorded, along with their relative abundance recorded as a percentage relative abundance of the total microbiome.
Change in Mammary Gland Microbiomes | Up to 26 months
  Investigators will examine the proportion of different bacteria taxa at each time point, and will use a marginalized two-part beta regression model to account for the compositional nature of the data. A list of all the microbiologic species will be recorded, along with their relative abundance recorded as a percentage relative abundance of the total microbiome.

CONTACTS AND LOCATIONS:
Overall Officials: Emily H Douglas, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No